CLINICAL TRIAL: NCT03436225
Title: Steroid Therapy in Acute Bronchiolitis A New Old Line of Therapy.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marina shohdy dous, Principal Investigator., Assiut University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Steroid in bronchiolitis.
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Bronchiolitis; Respiratory Syncytial Virus
Keywords: steroid therapy.
MeSH Terms: conditions — Bronchiolitis | interventions — dexamethasone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group one (Other): Group one will receive dexamethasone orally (0.15mg /kg / dose) twice daily for 3 to 5 days.
  Interventions: Drug: Dexamethasone orally.
- Group two (Other): Group two will receive dexamethasone parenteral (0.15mg /kg /dose) twice daily for 3 to 5 days.
  Interventions: Drug: Dexamethasone parenteral.
- Group three (Other): Group three will receive inhaled nebulized budesonide (1 mg/2ml) twice daily for 3 to 5 days.
  Interventions: Drug: Inhaled nebulized Budesonide.
- Group four (Other): Group four will receive symptomatic treatment in form of inhaled nebulized salbutamol(0.15mg/kg/ dose) daily every 6-8 hours.
  Interventions: Drug: Inhaled nebulized salbutamol.

INTERVENTIONS:
Drug: Dexamethasone orally. — Administered orally (0.15mg /kg / dose) twice daily for 3 to 5 days.
  Other Names: Apidone syrup.; Phenadone syrup.
  Arms: Group one
Drug: Dexamethasone parenteral. — Administered parenteral (0.15mg /kg / dose) twice daily for 3 to 5 days.
  Other Names: Fortecortin 8 mg /2 ml ampoule i.v /i.m injection .
  Arms: Group two
Drug: Inhaled nebulized Budesonide. — Administered for inhalation (1 mg/ 2ml) twice daily for 3 to 5 days.
  Other Names: Pulmicorte respules1 mg /2 ml.
  Arms: Group three
Drug: Inhaled nebulized salbutamol. — Administered for inhalation (0.15mg /kg / dose) daily every 6-8hrs
  Other Names: Farcoline respirator 0,5% solution.
  Arms: Group four

SUMMARY:
The aim of the present study is to evaluate the efficacy of steroid therapy and hospital stay in patients with acute bronchiolitis at assiut university children hospital.

DETAILED DESCRIPTION:
Bronchiolitis is an acute lower respiratory tract infection in early childhood.A subcommittee of the American Academy of Pediatrics (AAP) together with the European Respiratory Society (ERS) underlined that is a clinical diagnosis, recognized as "a constellation of clinical symptoms and signs including a viral upper respiratory prodrome followed by increased respiratory effort and wheezing in children less than 2 years of age".

Bronchiolitis is the common reason for hospitalization of children in many countries, challenging both economy, area and staffing in pediatric departments. A substantial proportion of children will experience at least one episode with bronchiolitis, and as much as 2-3% of all children will be hospitalized with bronchiolitis during their first year of life. Bronchiolitis is the most common medical reason for admission of children to intensive care units (ICU) particularly those with risk Factors will have a severe course of bronchiolitis, providing challenges regarding ventilation, fluid balance and general support This may be a particular challenge for ICUs without a specialized pediatric section.

Many respiratory viruses have been associated with acute viral bronchiolitis although Respiratory Syncytial Virus (RSV) remains the most common identified virus causing bronchiolitis, occurring in epidemics during winter months.The infection starts in the upper respiratory tract, spreading to the lower airways within few days.The inflammation in the bronchioles is characterized by a peri-bronchial infiltration of white blood cell types, mostly mono nuclear cells, and oedema of the submucosa and adventitia. Damage may occur by a direct viral injury to the respiratory airway epithelium, or indirectly by activating immune responses. Oedema, mucus secretion, and damage of airway epithelium with necrosis may cause partial or total airflow obstruction, distal air trapping, atelectasis and a ventilation perfusion mismatch leading to hypoxemia and increased work of breathing. Smooth-muscle constriction seems to play a minor role in the pathologic process of bronchiolitis.

Risk factors for bronchiolitis are male gender, a history of prematurity, young age, being born in relation to the RSV season, pre-existing disease such as broncho pulmonary- dysplasia , underlying chronic lung disease , neuromuscular disease, congenital heart- disease , exposure to environmental tobacco smoke , high parity, young maternal age, short duration/no breast feeding , maternal asthma and poor socioeconomic factors.

Bronchiolitis often starts with rhinorrhoea and fever, thereafter gradually increasing with signs of a lower respiratory tract infection including tachypnoea, wheezing and cough. Very young children, particularly those with a history of prematurity, may appear with apnea as their major symptom.Feeding problems are common.

On clinical examination, the major finding in the youngest children may be fine inspiratory crackles on auscultation, whereas high-pitched expiratory wheeze may be prominent in older children. By observation, the infants may have increased respiratory rate, chest movements, prolonged expiration, recessions, use of accessory muscles, cyanosis and decreased general condition.

No routine laboratory or radio graphic diagnostic tests for bronchiolitis except for pulse oxymetry , have been shown to have a substantial impact on the clinical course of bron- chiolitis , and recent guidelines and evidence-based reviews recommend that no diagnostic tests are used routinely.

The present study describes the efficacy of steroid therapy in patients with acute bronchiolitis. Theoretically, corticosteroid, an anti-inflammatory agent, should be helpful in the treatment of bronchiolitis because airway inflammation and edema are the main pathophysiologies. Recent evidence has shown elevation of interleukins and other inflammatory mediators in the respiratory tracts of children with acute bronchiolitis. Eosinophil cationic protein, implicated in the pathogenesis of asthma, was found to have a significant role in RSV bronchiolitis. Most of these mediators could be found during the period of virus replication.The clinical effect of dexamethasone, with a long half -life of 36-72 hr, may peak after 3-4 hr of treatment. Corticosteroids widely used in different routes in the treatment of acute bronchiolitis:

Dexamethasone injection used in hospitalized children with acute bronchiolitis showed significantly reduction in the mean respiratory distress duration, mean duration of oxygen therapy and the mean length of hospital stay.

Oral dexamethasone used in pediatric out patients with acute bronchiolitis produced demonstrable clinical improvement in the initial 4 hr of treatment and reduced the hospitalization rate.

Corticosteroid inhalation therapy used in RSV- bronchiolitis showed evidence of prolonged positive effects in reduction of the incidence of subsequent respiratory symptoms in the near future. However, the best and sufficient length of the treatment period, as well as the dose of the inhaled steroid, need to be determined..

Fluticasone propionate, a potent corticosteroid, has been demonstrated in vitro to inhibit virus-induced chemokine production by airway cells in patients infected with Respiratory Syncytial Virus. However, the inhibition was found to take at least 48 hr to reach its full effect.

ELIGIBILITY:
Inclusion Criteria:

1. Infants and young children aged from 3 months to 2 years with acute bronchiolitis.
2. Infants aged <12 months with respiratory rate over 60 breaths/min, childrens aged >12months with respiratory rate over 50 breaths/min.
3. Patients with an O2- saturation, breathing room air, under 95%.
4. Patients with apathy and/or refusal to eat.
5. Patients with normal white blood cell count for age.
6. Full term babies without chronic disease.

Exclusion Criteria:

1. Infants aged < 3 months, children aged >2 years
2. known or suspected asthma (by observing the good response to first dose of salbutamol nebulization especially among those with personal history of atopy).
3. Proven or suspected acute bacterial infection.
4. Presence of symptoms more than 7 days.
5. Previous treatment with corticosteroid by any route within 2 weeks.
6. Having a contra- indication to corticosteroid.
7. Severe cases requiring initial admission to intensive care unit with endotracheal intubation (in order to reduce confounding factors such as nosocomial infection or complication due to mechanical ventilation).
8. A previous history of intubation.
9. Premature babies (due to possible respiratory problems associated with prematurity).
10. Children with chronic cardiopulmonary diseases (Bronchopulmonary- dysplasia , Congenital Heart Disease and Cystic fibrosis)
11. Children with immunodeficiencies .
12. Children with neuromuscular disease.

Ages: 3 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Resolution of respiratory distress. | <7 days
  A total clinical score ≤ 3 and oxygen saturation ≥ 95 % at room air together with respiratory score of 0 or 1, a wheezing score of 0 or 1, and a retraction muscle score of 0 or 1

SECONDARY OUTCOMES:
Reduction of mean duration of symptoms. | <7 days
  Improvement of respiratory symptoms within fewer days .
Reduction of duration of oxygen therapy. | <7 days
  Reduction the need for more oxygen therapy .
Reduction of average Length of hospital stay. | <7 days
  Decrease Length of hospital stay.

REFERENCES:
- [Background] Schimmer BP, Parker KL. Adrenocorticotropic hormone; adrenocortical steroids and their synthetic analogs; inhibitor of the synthesis and actions of adrenocortical hormones. In: Hardman JG, Limbird LE, Molinoff PB, Ruddon RW, Gilman AG,editors. Goodman & Gilman's the pharmacological basis of therapeutics, 9th edition. New York: McGraw-Hill; 1996.pp 1459-1485.
- [Background] GOODWIN A. An uncontrolled assessment of nebulized budesonide in the treatment of acute bronchiolitis. Br J Clin Res 1995: 6: 113±9.
- [Result] Nagakumar P, Doull I. Current therapy for bronchiolitis. Arch Dis Child. 2012 Sep;97(9):827-30. doi: 10.1136/archdischild-2011-301579. Epub 2012 Jun 25. PMID 22734014
- [Result] American Academy of Pediatrics Subcommittee on Diagnosis and Management of Bronchiolitis. Diagnosis and management of bronchiolitis. Pediatrics. 2006 Oct;118(4):1774-93. doi: 10.1542/peds.2006-2223. PMID 17015575
- [Result] Stockman LJ, Curns AT, Anderson LJ, Fischer-Langley G. Respiratory syncytial virus-associated hospitalizations among infants and young children in the United States, 1997-2006. Pediatr Infect Dis J. 2012 Jan;31(1):5-9. doi: 10.1097/INF.0b013e31822e68e6. PMID 21817948
- [Result] Choi J, Lee GL. Common pediatric respiratory emergencies. Emerg Med Clin North Am. 2012 May;30(2):529-63, x. doi: 10.1016/j.emc.2011.10.009. Epub 2011 Dec 17. PMID 22487117
- [Result] Zorc JJ, Hall CB. Bronchiolitis: recent evidence on diagnosis and management. Pediatrics. 2010 Feb;125(2):342-9. doi: 10.1542/peds.2009-2092. Epub 2010 Jan 25. PMID 20100768
- [Result] Wainwright C. Acute viral bronchiolitis in children- a very common condition with few therapeutic options. Paediatr Respir Rev. 2010 Mar;11(1):39-45; quiz 45. doi: 10.1016/j.prrv.2009.10.001. Epub 2009 Nov 26. PMID 20113991
- [Result] Carroll KN, Gebretsadik T, Griffin MR, Wu P, Dupont WD, Mitchel EF, Enriquez R, Hartert TV. Increasing burden and risk factors for bronchiolitis-related medical visits in infants enrolled in a state health care insurance plan. Pediatrics. 2008 Jul;122(1):58-64. doi: 10.1542/peds.2007-2087. PMID 18595987
- [Result] Murray J, Bottle A, Sharland M, Modi N, Aylin P, Majeed A, Saxena S; Medicines for Neonates Investigator Group. Risk factors for hospital admission with RSV bronchiolitis in England: a population-based birth cohort study. PLoS One. 2014 Feb 26;9(2):e89186. doi: 10.1371/journal.pone.0089186. eCollection 2014. PMID 24586581
- [Result] Bordley WC, Viswanathan M, King VJ, Sutton SF, Jackman AM, Sterling L, Lohr KN. Diagnosis and testing in bronchiolitis: a systematic review. Arch Pediatr Adolesc Med. 2004 Feb;158(2):119-26. doi: 10.1001/archpedi.158.2.119. PMID 14757603
- [Result] Sheeran P, Jafri H, Carubelli C, Saavedra J, Johnson C, Krisher K, Sanchez PJ, Ramilo O. Elevated cytokine concentrations in the nasopharyngeal and tracheal secretions of children with respiratory syncytial virus disease. Pediatr Infect Dis J. 1999 Feb;18(2):115-22. doi: 10.1097/00006454-199902000-00007. PMID 10048682
- [Result] Noah TL, Becker S. Respiratory syncytial virus-induced cytokine production by a human bronchial epithelial cell line. Am J Physiol. 1993 Nov;265(5 Pt 1):L472-8. doi: 10.1152/ajplung.1993.265.5.L472. PMID 8238534
- [Result] Garofalo R, Kimpen JL, Welliver RC, Ogra PL. Eosinophil degranulation in the respiratory tract during naturally acquired respiratory syncytial virus infection. J Pediatr. 1992 Jan;120(1):28-32. doi: 10.1016/s0022-3476(05)80592-x. PMID 1731020
- [Result] Volovitz B, Faden H, Ogra PL. Release of leukotriene C4 in respiratory tract during acute viral infection. J Pediatr. 1988 Feb;112(2):218-22. doi: 10.1016/s0022-3476(88)80058-1. PMID 3339502
- [Result] Roosevelt G, Sheehan K, Grupp-Phelan J, Tanz RR, Listernick R. Dexamethasone in bronchiolitis: a randomised controlled trial. Lancet. 1996 Aug 3;348(9023):292-5. doi: 10.1016/s0140-6736(96)02285-4. PMID 8709687
- [Result] De Boeck K, Van der Aa N, Van Lierde S, Corbeel L, Eeckels R. Respiratory syncytial virus bronchiolitis: a double-blind dexamethasone efficacy study. J Pediatr. 1997 Dec;131(6):919-21. doi: 10.1016/s0022-3476(97)70044-1. PMID 9427901
- [Result] Klassen TP, Sutcliffe T, Watters LK, Wells GA, Allen UD, Li MM. Dexamethasone in salbutamol-treated inpatients with acute bronchiolitis: a randomized, controlled trial. J Pediatr. 1997 Feb;130(2):191-6. doi: 10.1016/s0022-3476(97)70342-1. PMID 9042119
- [Result] Berger I, Argaman Z, Schwartz SB, Segal E, Kiderman A, Branski D, Kerem E. Efficacy of corticosteroids in acute bronchiolitis: short-term and long-term follow-up. Pediatr Pulmonol. 1998 Sep;26(3):162-6. doi: 10.1002/(sici)1099-0496(199809)26:33.0.co;2-n. PMID 9773910
- [Result] Schuh S, Coates AL, Binnie R, Allin T, Goia C, Corey M, Dick PT. Efficacy of oral dexamethasone in outpatients with acute bronchiolitis. J Pediatr. 2002 Jan;140(1):27-32. doi: 10.1067/mpd.2002.120271. PMID 11815760
- [Result] Maayan C, Itzhaki T, Bar-Yishay E, Gross S, Tal A, Godfrey S. The functional response of infants with persistent wheezing to nebulized beclomethasone dipropionate. Pediatr Pulmonol. 1986 Jan-Feb;2(1):9-14. doi: 10.1002/ppul.1950020106. PMID 3513105
- [Result] Reijonen T, Korppi M, Kuikka L, Remes K. Anti-inflammatory therapy reduces wheezing after bronchiolitis. Arch Pediatr Adolesc Med. 1996 May;150(5):512-7. doi: 10.1001/archpedi.1996.02170300066013. PMID 8620234
- [Result] Carlsen KH, Leegaard J, Larsen S, Orstavik I. Nebulised beclomethasone dipropionate in recurrent obstructive episodes after acute bronchiolitis. Arch Dis Child. 1988 Dec;63(12):1428-33. doi: 10.1136/adc.63.12.1428. PMID 3069051
- [Result] Noah TL, Wortman IA, Becker S. The effect of fluticasone propionate on respiratory syncytial virus-induced chemokine release by a human bronchial epithelial cell line. Immunopharmacology. 1998 Jun;39(3):193-9. doi: 10.1016/s0162-3109(98)00017-4. PMID 9754905
- [Result] Tal A, Bavilski C, Yohai D, Bearman JE, Gorodischer R, Moses SW. Dexamethasone and salbutamol in the treatment of acute wheezing in infants. Pediatrics. 1983 Jan;71(1):13-8. PMID 6129609